CLINICAL TRIAL: NCT01124500
Title: Efficacy and Safety of Transdermal Methylphenidate for Cancer-Related Fatigue
Brief Title: Transdermal Methylphenidate for Cancer-Related Fatigue
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Natalie Moryl, MD, Memorial Sloan-Kettering Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10-020
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Last update posted 2010-08-26 (Estimated); Status verified 2010-08

CONDITIONS: Head and Neck Cancer
Keywords: methylphenidate; transdermal patch; placebo; fatigue; 10-020
MeSH Terms: conditions — Head and Neck Neoplasms; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- methylphenidate via transdermal patch compared to placebo (Experimental): The proposed study is a within-subject, cross-over, randomized and double-blinded pilot trial, designed to evaluate the efficacy and feasibility of sustained-release, long-acting methylphenidate via transdermal patch compared to placebo in fatigued patients with Head and Neck malignancies
  Interventions: Drug: methylphenidate via transdermal patch compared to placebo

INTERVENTIONS:
Drug: methylphenidate via transdermal patch compared to placebo — The participants will start with a 10mg MPH patch on day -4, the 1st day of the titration period. This will be increased up to 20mg over 4-day titration period as needed and tolerated, and continued on the optimal dose. Subjects will be seen on day 1 of the double-blind part of the study at a patient education room or the Dr.'s office and receive 10 identical patches including 5 MPH and 5 placebo patches that will be randomly assigned over the 10-day course. The patch will be placed at 9am and removed at 4pm daily for 10 days. During the 10 days, each subject will be monitored for continuous 240 hours by actigraphy based activity monitors to follow activity levels and energy expenditure.

SUMMARY:
The purpose of this study is to compare the effects, good and/or bad, of the Methylphenidate patch and a placebo patch (a patch that contains no medicine) on patients and their fatigue caused by cancer or by cancer treatment. The Methylphenidate patch contains a medication that is known to increase alertness and wakefulness. Oral methylphenidate has been used in the past to treat cancer related fatigue and is often used to treat unusual sleepiness. But this is the first time that the patch form is offered to try treating cancer fatigue in patients who cannot always swallow tablets.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of head and neck cancer who underwent combined modality treatment with curative intent
* Has not undergone cancer treatment in the last 4 weeks
* Is 21 years of age or older
* Fatigue scale score of 4 or higher
* Is able to understand English, through written and verbal communication
* In the judgment of the consenting professional, is able to provide informed consent
* Physically able to present for follow-up appointments at outpatient Radiation Oncology or Pain & Palliative Care clinics
* Probable life expectancy of more than 6 months

Exclusion Criteria:

* Pulmonary or cardiovascular failure, seizure disorder, sleep disorder, mental impairment, psychiatric disorder, or pregnancy
* Has known sensitivity or allergies to methylphenidate
* Receiving concurrent treatment with a psychostimulant
* Hospitalized patients
* Evidence of impaired hepatic or renal function (hyperbilirubinemia, greater than two fold elevation of transaminases; >40mg/dl BUN or >1.5mg/dl Cr )
* Anemia ( hemoglobin <10mg/dl)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
To investigate the efficacy of sustained-release, transdermal methylphenidate compared to a placebo. | for 10 days
  In reducing fatigue, increasing activity levels, and sustaining steady wakefulness throughout the day. The outcome measure will be BFI and ESS based self-reporting of the reduction of numeric rating scale on fatigue level and sleepiness, combined with objective measurement of increased activity intensity scores monitored by actigraphy.
To evaluate the possible side effects of a methylphenidate patch. | for 10 days
  In adult head and neck cancer patients with fatigue.

SECONDARY OUTCOMES:
To evaluate the feasibility of accelerometry-based objective outcome measures to assess improved activity levels and energy expenditure of cancer patients. | for 10 days
  To evaluate the feasibility of accelerometry-based objective outcome measures to assess improved activity levels and energy expenditure, will be evaluated by examining the patients' rating of their comfort while wearing the actigraphy device and of how willing they would be to wear the device for a future study.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Moryl, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org